CLINICAL TRIAL: NCT06793267
Title: Ultrasonoraphic Asessment of Metoclopramide Effect on Gastric Volume in Urgent Surgical Trauma Pediateric Patients. Randomozed Controlled Double Blind Study.
Brief Title: Ultrasound Assessment of Metoclopramide's Effect on Stomach Volume in Urgent Pediatric Trauma Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Ahmed Ali Hamed, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USAMEGVUSTP
Record Dates: First submitted 2025-01-15; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Gastric Volume
MeSH Terms: interventions — Metoclopramide; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group1 (Active Comparator): patients will receive 0.15mg/kg metoclopramide intravenously diluted in 2 ml.
  Interventions: Drug: Metoclopramide (Maxolon)
- Group 2 (Placebo Comparator): Participants will receive a placebo in the form of 2 ml of normal saline administered intravenously.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Metoclopramide (Maxolon) — Participants will receive 0.15 mg/kg of metoclopramide administered intravenously. The drug will be diluted in 2 ml of solution prior to administration.
  Arms: Group1
Drug: Saline — patients will recive normal saline 0.9% 2ml intravenous
  Arms: Group 2

SUMMARY:
assess the efficacy of metoclopramide in reducing the gastric contents and volume in pediatric trauma prepared for urgent surgical interventions.

DETAILED DESCRIPTION:
Gastric volume is a critical consideration in pediatric patients undergoing urgent surgical procedures, particularly in trauma cases where rapid sequence induction is required to minimize the risk of aspiration. Point-of-care gastric ultrasonography (gastric PocUs) allows evaluation of the volume and type of stomach contents. Previous studies have reported that gastric contents and volume measured using gastric PoCUS are significantly correlated with cross-sectional antral area. as a result, bedside gastric PocUs is considered a reliable and reproducible technique. gastric PocUs scan can distinguish an empty stomach from a full stomach based on qualitative results by distinguishing the physical properties of gastric fluid. The presence of thick fluid and solid contents indicate a full stomach.in contrast, the presence of clear gastric fluid is normal in healthy, fasted individuals at low risk of aspiration. as a result, assessing the volume of clear fluid in the stomach may have utility in identifying high stomach volumes that are incompatible with the fasting state.

Metoclopramide is a prokinetic chlorobenzamide derivative that accelerates gastric emptying and reduces gastric volume. Metoclopramide can be safely used preoperatively prior to cesarean section (cs). Metoclopramide has been extensively studied as a premedication for abdominal surgery, particularly in obstetric populations. Due to favorable effect of reducing gastric fluid volume, metoclopramide is commonly used to reduce the risk of aspiration pneumonia during surgery. Metoclopramide reportedly has synergistic dual activity in parturient women; an antiemetic effect on the chemoreceptor trigger zone and peripheral activity in increasing the tone of the lower esophageal sphincter and decreasing the time required for gastric emptying. the mortality of aspiration pneumonia-related is reportedly as high as 5%, with aspiration pneumonia responsible for up to 9% of all anesthesia-related deaths. Metoclopramide is well known for its ability to enhance gastric emptying however, to the best of our knowledge, the effectiveness of metoclopramide in enhancing gastric emptying has yet to be evaluated with ultrasonography in preoperative settings, particularly in urgent pediatric trauma.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric urgent trauma

Exclusion Criteria:

* Guardian' refusal.
* Presence of head trauma.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
ultrasonographic assessment of the effect of metoclopramide on morphology of the gastric antrum | baseline
  Ultrasonographic evaluation was performed to study the impact of metoclopramide on the morphology of the gastric antrum. The cross-sectional area (CSA) of the antrum was calculated using the Bolondi et al. method with the formula:Antral CSA = π (AP × CC) / 4

SECONDARY OUTCOMES:
effect of metoclopramide on gastric grading was assessed using a three-point grading systems | baseline
  The effect of metoclopramide on gastric grading was evaluated using a three-point grading system as follows:
  G-0: The antrum is flat and empty in both supine and right lateral positions (RLP).
  G-1: The antrum contains fluid in the right lateral position but is empty in the supine position.
  G-2: The antrum contains fluid in both supine and right lateral positions.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bolondi L, Bortolotti M, Santi V, Calletti T, Gaiani S, Labo G. Measurement of gastric emptying time by real-time ultrasonography. Gastroenterology. 1985 Oct;89(4):752-9. doi: 10.1016/0016-5085(85)90569-4. PMID 3896910
- [Background] Howard FA, Sharp DS. Effect of metoclopramide on gastric emptying during labour. Br Med J. 1973 Feb 24;1(5851):446-8. PMID 4689832
- [Background] Adelhoj B, Petring OU, Pedersen NO, Andersen RD, Busch P, Vestergard AS. Metoclopramide given pre-operatively empties the stomach. Acta Anaesthesiol Scand. 1985 Apr;29(3):322-5. doi: 10.1111/j.1399-6576.1985.tb02208.x. PMID 3993321
- [Background] simeneh endalew EN, gebremedhn eg, gebreegzi aH, gebreegzi AH, Kassahun HG, Kassa AA, et al. effectiveness of intravenous metoclopramide prophylaxis on the reduction of intraoperative and early postoperative nausea and vomiting after emergency caesarean section under spinal anaesthesia. J anesth clin res 2018;09:2.
- [Background] O'Sullivan G, Sear JW, Bullingham RE, Carrie LE. The effect of magnesium trisilicate mixture, metoclopramide and ranitidine on gastric pH, volume and serum gastrin. Anaesthesia. 1985 Mar;40(3):246-53. doi: 10.1111/j.1365-2044.1985.tb10750.x. PMID 2986474
- [Background] Paranjothy S, Griffiths JD, Broughton HK, Gyte GM, Brown HC, Thomas J. Interventions at caesarean section for reducing the risk of aspiration pneumonitis. Cochrane Database Syst Rev. 2014 Feb 5;2014(2):CD004943. doi: 10.1002/14651858.CD004943.pub4. PMID 24497372
- [Background] Kruisselbrink R, Gharapetian A, Chaparro LE, Ami N, Richler D, Chan VWS, Perlas A. Diagnostic Accuracy of Point-of-Care Gastric Ultrasound. Anesth Analg. 2019 Jan;128(1):89-95. doi: 10.1213/ANE.0000000000003372. PMID 29624530
- [Background] Van de Putte P, Perlas A. Ultrasound assessment of gastric content and volume. Br J Anaesth. 2014 Jul;113(1):12-22. doi: 10.1093/bja/aeu151. Epub 2014 Jun 3. PMID 24893784